CLINICAL TRIAL: NCT00027716
Title: A Multi-Institutional, Open-Label, Two-Group, Phase II Study of PS-341 (LDP-341, NSC #681239) in Patients With Advanced or Metastatic Sarcoma
Brief Title: Bortezomib in Treating Patients With Advanced or Metastatic Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 01-073; CDR0000069060 (Registry Identifier: PDQ (Physician Data Query)); NCI-1757
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Sarcoma
Keywords: metastatic osteosarcoma; recurrent adult soft tissue sarcoma; recurrent osteosarcoma; adult rhabdomyosarcoma; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Osteosarcoma; Rhabdomyosarcoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer by blocking the enzymes necessary for tumor cell growth.

PURPOSE: Phase II trial to study the effectiveness of bortezomib in treating patients who have advanced or metastatic sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with advanced or metastatic sarcoma treated with bortezomib.
* Correlate levels of cyclins D1, E, p21 (WAF1), p27 (Kip1), mdm^2, p53, and Ki67 with response in patients treated with this drug.

OUTLINE: This is an open-label, multicenter study. Patients are stratified according to disease (stratum I: soft tissue sarcoma not specified in stratum II, osteogenic sarcoma arising from soft tissues, or gastrointestinal stromal tumor vs stratum II: Ewing's sarcoma of soft tissue or bone, rhabdomyosarcoma, or osteogenic sarcoma of bone). (Stratum I closed to accrual as of 10/17/03.)

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 21-41 patients will be accrued for stratum I within 5-11 months and 21-41 patients will be accrued for stratum II within 10.5-22 months. (Stratum I closed to accrual as of 10/17/03.)

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed sarcoma
* Soft tissue metastasis or locally recurrent disease
* Stratum I (closed to accrual as of 10/17/03):

  * Soft tissue sarcoma not specified in stratum II
  * Osteogenic sarcoma arising from soft tissue or gastrointestinal stromal tumor (GIST)
* Stratum II:

  * Ewing's sarcoma of soft tissue or bone (if measurable soft tissue metastasis is present)
  * Rhabdomyosarcoma
  * Osteogenic sarcoma of bone (if measurable soft tissue metastasis is present)
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
* Disease progression within the past 3 months
* No prior or active known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 80-100% OR
* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST/ALT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No peripheral vascular disease requiring surgical management
* No history of congestive heart failure even if it is medically controlled
* No angina pectoris even if it is medically controlled
* No myocardial infarction within the past year
* No cardiac arrhythmias
* No prior cerebrovascular event
* No prior transient ischemic attack
* No EKG evidence of acute ischemia or conduction abnormality (e.g., bifascicular block [left anterior hemiblock in the presence of right bundle branch block] or second or third degree atrioventricular block)
* No history of orthostatic hypotension

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reaction to compounds of similar chemical or biological composition to study drug
* No other uncontrolled concurrent illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other malignancy within the past 5 years except adequately treated basal cell skin cancer or carcinoma in situ of the cervix
* No symptomatic peripheral neuropathy greater than grade 1

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered
* No concurrent biological or immunological agents

Chemotherapy:

* Stratum I (closed to accrual as of 10/17/03):

  * At least 1 year since prior chemotherapy in the adjuvant or neoadjuvant setting
  * No other prior chemotherapy
* Stratum II:

  * No more than 1 prior chemotherapy regimen
* No concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* Prior imatinib mesylate for GIST (stratum I closed to accrual as of 10/17/03) allowed
* No other concurrent investigational agents
* No concurrent commercial anticancer agents or therapies
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-10; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Maki, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Chicago Cancer Research Center, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Abramson Cancer Center at University of Pennsylvania Medical Center, Philadelphia, Pennsylvania